CLINICAL TRIAL: NCT02924753
Title: The Safety and Efficacy of CART-19 Cells in Relapse and Refractory Patients With CD19+ B-cell Acute Lymphoblastic Leukemia.
Brief Title: The Safety and Efficacy of CART-19 Cells in B-cell Acute Lymphoblastic Leukemia (B-ALL).
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: The Beijing Pregene Science and Technology Company, Ltd. (Industry)
Responsible Party: Principal Investigator, Yongping Song, director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH080
Record Dates: First submitted 2016-09-29; First posted 2016-10-05 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CART-19 (Experimental): patients will receive a pre-conditioning with cyclophosphamide and fludarabine before infusion of CART-19 cells. The CART-19 cells are to be administered on day0,day1,day2.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: CART-19 cells

INTERVENTIONS:
Drug: Cyclophosphamide — patients will receive a standard pre-conditioning regime with cyclophosphamide 0.8-1.0g/m2/day IV for 2 days(Day-5 to day-4).
Drug: Fludarabine — Fludarabine 25mg/m2/day IV for 3 days (Day-5 to day-3).
Biological: CART-19 cells — CART-19 cells will be administered using a split dose on day0(10%), 1(30%), and 2(60%) after completion of the chemotherapy.
  Other Names: CD19 specific Chimeric Antigen Receptor T-cells

SUMMARY:
This is a study for patients who have been previously treated for B-ALL. The purpose of this study is to determine the safety and feasibility of CART-19 cells to the patients with relapsed and refractory CD19+ B-ALL.

DETAILED DESCRIPTION:
Subjects will be staged and the suitability of their T cells for CART-19 manufacturing will be determined at entry phase,. Subjects will be collected large numbers of peripheral blood mononuclear cells (PBMC) for CART-19 manufacturing. The T cells will be purified from the PBMC, transduced with CART-19 lentiviral vector, expanded in vitro and then administered to subjects.

Subjects will have blood tests to assess safety and efficacy, and persistence of the CART-19 cells at regular intervals through four weeks after their last infusion of the study. Following the 6 months of intensive follow-up, subjects will be evaluated quarterly for two years with a physical examination, blood tests, bone marrow aspirate, minimal residual disease (MRD) and persistence of CART-19. Following this evaluation, subjects will be evaluated health problems every year for an additional thirteen years.

ELIGIBILITY:
Inclusion Criteria:

1. 4 years to 70 years, expected survival > 3 months
2. CD19 positive B-cell acute lymphoblastic leukemia
3. Karnofsky Performance Status (KPS) >70
4. Relapsed after allogeneic or autologous stem cell transplantation (SCT);
5. Cardiac function: 1-2 levels; Liver: TBIL≤3 Upper Limit of Normal (ULN)，aspartate aminotransferase (AST) ≤2.5 ULN，ALT ≤2.5 ULN; kidney: Cr≤1.25 ULN; bone marrow: White Blood Cell (WBC) ≥ 3.0×109/L, Hb ≥90 g/L, Platelet (PLT) ≥ 80×109/L）
6. No serious allergic constitution
7. No other serous diseases that conflicts with the clinical program
8. No other cancer history
9. No serious mental disorder
10. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. Pregnant or lactating women; (female participants of reproductive potential must have a negative serum or urine pregnancy test)
2. Uncontrolled active infection, HIV infection, syphilis serology reaction positive
3. Active hepatitis B or hepatitis C infection
4. Recent or current use of glucocorticoid or other immunosuppressor
5. With severe cardiac, liver, renal insufficiency, diabetes and other diseases
6. Transaminase >2.5 ULN, Bilirubin >3 ULN，Creatinine>1.25 ULN
7. Participate in other clinical research in the past three months; previously treatment with any gene therapy products
8. Researchers think of that does not fit to participate in the study, or other cases that affect the clinical trial results

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07-18 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
safety as assessed by the occurrence of study related adverse events. | 6 months
  monitor the occurrence of study related adverse events.

SECONDARY OUTCOMES:
efficacy | 2 years
  anti-tumor activity of CART-19 cells will be determined in a follow-on study
duration of CART-19 | 2 years
  Determine duration of in vivo survival of CART-19 cells.

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China